CLINICAL TRIAL: NCT05509374
Title: Phase II, Single-arm Trial of Carfilzomib, Pomalidomide, and Dexamethasone for Myeloma Patients Who Had Relapsed or Progressed After Carfilzomib, Lenalidomide, and Dexamethasone
Brief Title: Phase II Study of Carfilzomib, Pomalidomide, and Dexamethasone for Myeloma Patients Who Had Relapsed or Progressed After Carfilzomib, Lenalidomide, and Dexamethasone
Acronym: KMM2002
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kihyun Kim, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC-2021-03-147
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A study of carfilzomib, pomalidomide and dexamethasone administration after KRd administration (Experimental): Patients with RRMM who progressed after receiving lenalidomide monotherapy for at least 6 months after administration of KRd will receive KPD therapy every 4 weeks until disease progression.
  Interventions: Drug: Carfilzomib 56 MG [Kyprolis]; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib 56 MG [Kyprolis] — Carfilzomib 56 mg/m2 (Day1, 8, 15) (Cycle1 Day1, 20 mg/m2)
Drug: Pomalidomide — Pomalidomide 4 mg per os (Day1-21)
Drug: Dexamethasone — Dexamethasone 40 mg (D1, 8, 15, 22) (20 mg for patients ≥ 75 years old)

SUMMARY:
The purpose of this study is to evaluate the evaluate the efficacy and safety of administering a combination of carfilzomib, pomalidomide, and dexamethasone in patients with relapsed or advanced multiple myeloma after carfilzomib, lenalidomide, and dexamethasone therapy.

DETAILED DESCRIPTION:
This study is a phase 2 study in which patients with RRMM under 80 years of age who have been treated with lenalidomide monotherapy for at least 6 months after KRd combination therapy will receive carfilzomib, pomalidomide, and dexamethasone combination therapy.

A total of 33 participants are recruited.

KPd will be administered until progressive disease or unacceptable toxicities.

Participants who discontinued treatment will be followed up for disease status and survival at 2-month intervals.

Responses are assessed using the International Myeloma Working Group (IMWG) response criteria and the safety profile is described using NCI-CTCAE v5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 20 to 80 years-old
2. Relapse or progression of multiple myeloma after treatment of carfilzomib/lenalidomide/dexamethasone (KRd)
3. KRd treatment 12 cycles or more and lenalidomide maintenance for at least 6 months or KRd 4-6 cycles followed by ASCT and lenalidomide maintenance for at least 6 months
4. Measurable disease

   * Serum M-protein ≥ 1 g/dL (10 g/L)
   * Urine M-protein ≥ 200 mg/24 hr
   * Serum FLC assay: difference of FLC ≥ 10 mg/dL (100 mg/L) provided serum FLC ratio is abnormal (KL ratio < 0.26 or > 1.65) if Serum EP or urine EP is not measurable
5. Adequate organ functions

   * Absolute Neutrophil Count (ANC) ≥ 1.0 x 109/L
   * Platelets ≥ 50 x 109/L (≥ 30 x 109/L if myeloma involvement is > 50% in the bone marrow)
   * Hemoglobin ≥ 8.0 g/dL
   * Creatinine clearance ≥ 30 mL/minute or Serum Cr <3.0 g/dL
   * Serum Bilirubin ≤ 1.5 x ULN
   * AST and ALT ≤ 3 x ULN
6. Eastern Cooperative Oncology Group performance scale 0~2
7. Life expectancy longer than 3 months
8. Written informed consent
9. Prior therapy with bortezomib
10. Patients who meet the following criteria

    * If a woman of childbearing age

      * Women who are willing to use two reliable methods of contraception from 4 weeks prior to administration of study drug, while receiving, temporarily suspending administration, and 4 weeks after administration of the study drug.
      * Women who have a negative pregnancy test with a minimum sensitivity of 25 IU/mL under medical management
    * For men Men who agree to abstain from absolute abstinence or use a proper method of contraception for the entire duration of treatment and 28 days after the last dose

      * Women of childbearing age Women who have not undergone hysterectomy or bilateral oophorectomy, women who have not undergone spontaneous menopause for at least 24 consecutive months (i.e., menstruate at any time during the last 24 months. However, amenorrhea after chemotherapy does not exclude the possibility of pregnancy).
      * Proper method of contraception
    * Very effective way Intrauterine device, hormone therapy (hormone implant, intrauterine system releasing levonorgestrel, medroxyprogesterone acetate depot injection, tablets containing progesterone to inhibit ovulation), tubal ligation, varicose veins in men
    * Effective way Men's condom use, diaphragm method, cervical cap

Exclusion Criteria:

1. Grade 3~4 non-hematologic toxicity by carfilzomib during the previous carfilzomib treatment
2. Prior therapy with pomalidomide
3. Hypersensitivity to thalidomide or lenalidomide
4. Previous refractoriness to carfilzomib according to the IMWG criteria
5. Myocardial infarct within 6 months, heart failure of NYHA Class III~IV, uncontrolled ventricular arrhythmia, severe coronary arterial obstructive disease
6. Active infection with 14 days prior to treatment
7. Uncontrolled hypertension (Defined as an average systolic blood pressure >= 160 mmHg or diastolic >= 100 mmHg) or diabetes (HbA1c > 7.0%)
8. HIV, HBV, HCV infection (exception if adequately controlled HBV (undetectable HBV DNA (< 20 IU/mL or concurrent use of an anti-viral agent), HCV)
9. Severe or uncontrolled medical conditions, laboratory abnormalities, or psychiatric disorders that may preclude the participation of the study by the physician's discretion
10. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
11. Diagnosis of other malignant disease other than myeloma within 5 year. Exceptions are properly treated non-melanomatous skin cancers, cervical intraepithelial neoplasia, prostate cancer that do not require treatment, or properly excised well-differentiated thyroid cancers.
12. Pregnant or nursing women
13. Waldenstroem's macroglobulinemia, POEMS syndrome, or plasma cell leukemia, light chain amyloidosis
14. LV ejection fraction < 40%

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | assessed for approximately 3 years after administration
  percentage of patients who achieve at least partial response

SECONDARY OUTCOMES:
Complete response rate | assessed for approximately 3 years after administration
  percentage of patients who achieve complete response
Progression free survival rate | assessed for approximately 3 years after administration
  percentage of patients who are disease free or alive
Overall survival | assessed for approximately 3 years after administration
  from the time of written consent to the time of death or last follow-up
Duration of response | assessed for approximately 3 years after administration
  from the time of achieving at least partial response to the time of progressive disease
Time to response | assessed for approximately 3 years after administration
  from the time of written consent to the time of achieving at least partial response
Incidence of treatment-emergent adverse events | assessed for approximately 3 years after administration
  Safety profiles of carfilzomib, pomalidomide, and dexamethasone for myeloma patients who had relapsed or progressed
Minimal residual disease negativity | up to 3 years
  The specimen is bone marrow aspirate, and it should be free of clonal plasma cells by examination by the NGF (next-generation flow) method. At this time, the test should be performed according to the EuroFlow standard operation procedure for MRD detection in MM, and the minimum sensitivity should be10 to the 5th power or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Kihyun Kim, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No